CLINICAL TRIAL: NCT03491748
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Oral ETX0282 Administered in Healthy Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics (PK, the Measure of How the Human Body Processes a Substance) of ETX0282 When Administered Orally to Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Entasis Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CS0282-2017-0001; 1010452 (Other: INC Research)
Record Dates: First submitted 2018-03-23; First posted 2018-04-09 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; ETX0282; Single Ascending Dose; Multiple Ascending Doses; ETX1317; Cefpodoxime Proxetil; Cefpodoxime; Enterobacteriaceae Infections
MeSH Terms: conditions — Enterobacteriaceae Infections | interventions — Cefpodoxime Proxetil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Part A (SAD): Cohort 1, 100 mg ETX0282/Placebo (Experimental): Part A of the study will explore the safety, tolerability, and pharmacokinetics (PK) of a single ascending dose (SAD) of oral ETX0282. Participants will be treated with a single oral dose of 100 milligrams (mg) ETX0282 or placebo in a fasted state. They will be confined to the Study Unit from Day -1 and discharged following collection of the 72-hour postdose assessments (Day 4).
  Interventions: Drug: ETX0282; Drug: Placebo
- Part A (SAD): Cohort 2, 200 mg ETX0282/Placebo (Experimental): Part A of the study will explore the safety, tolerability, and PK of a SAD of oral ETX0282. Participants will be treated with a single oral dose of 200 mg ETX0282 or placebo in a fasted state. They will be confined to the Study Unit from Day -1 and discharged following collection of the 72-hour postdose assessments (Day 4).
  Interventions: Drug: ETX0282; Drug: Placebo
- Part A (SAD): Cohort 3, 400 mg ETX0282/Placebo (Experimental): Part A of the study will explore the safety, tolerability, and PK of a SAD of oral ETX0282. Participants will be treated with a single oral dose of 400 mg ETX0282 or placebo in a fasted state. They will be confined to the Study Unit from Day -1 and discharged following collection of the 72-hour postdose assessments (Day 4).
  Interventions: Drug: ETX0282; Drug: Placebo
- Part A (SAD): Cohort 4, 800 mg ETX0282/Placebo (Experimental): Part A of the study will explore the safety, tolerability, and PK of a SAD of oral ETX0282. Participants will be treated with a single oral dose of 800 mg ETX0282 or placebo in a fasted state. They will be confined to the Study Unit from Day -1 and discharged following collection of the 72-hour postdose assessments (Day 4).
  Interventions: Drug: ETX0282; Drug: Placebo
- Part A (SAD): Cohort 5, 600 mg ETX0282/Placebo (Experimental): Part A of the study will explore the safety, tolerability, and PK of a SAD of oral ETX0282. Participants will be treated with a single oral dose of 600 mg ETX0282 or placebo in a fasted state. They will be confined to the Study Unit from Day -1 and discharged following collection of the 72-hour postdose assessments (Day 4).
  Interventions: Drug: ETX0282; Drug: Placebo
- Part A (SAD): Cohort 6 (Elderly), 300 mg ETX0282/Placebo (Experimental): Part A of the study will explore the safety, tolerability, and PK of a SAD of oral ETX0282. Elderly participants (aged 65 years or older) will be treated with a single oral dose of 300 mg ETX0282 or placebo in a fasted state. They will be confined to the Study Unit from Day -1 and discharged following collection of the 72-hour postdose assessments (Day 4).
  Interventions: Drug: ETX0282; Drug: Placebo
- Part B (Food Effect): Cohort 7, 100 mg ETX0282/Placebo (Experimental): Part B of the study will explore the effect of food on oral ETX0282. Participants will be treated with a single oral dose of 100 mg ETX0282 or placebo (Day 1) while fasted and with a single oral dose of 100 mg ETX0282 or placebo (Day 4) with a high-fat meal. They will be confined to the Study Unit from Day -1 and discharged following collection of the 72-hour post fed state dose assessments (Day 7).
  Interventions: Drug: ETX0282; Drug: Placebo
- Part C (MAD): Cohort 9, 200 mg ETX0282/Placebo (Experimental): Part C of the study will explore the safety, tolerability, and PK of MAD of oral ETX0282. Part C will be administered in a fed state. Participants will be treated with a single oral dose of 200 mg ETX0282 or placebo on the morning of Day 1, and will then be dosed three times a day (TID) beginning on the morning of Day 2 (i.e., 24 hours after the Day 1 dose) through Day 7. Participants will be treated with a single oral dose of 200 mg ETX0282 or placebo on the morning of Day 8. They will be confined to the Study Unit from Day -1 and discharged following collection of the 72-hour post Day 8 dose assessments (Day 11).
  Interventions: Drug: ETX0282; Drug: Placebo
- Part C (MAD): Cohort 10, 200 mg ETX0282/Placebo (Experimental): Part C of the study will explore the safety, tolerability, and PK of MAD of oral ETX0282. Part C will be administered in a fed state. Participants will be treated with a single oral dose of 200 mg ETX0282 or placebo on the morning of Day 1, and will then be dosed TID beginning on the morning of Day 2 (i.e., 24 hours after the Day 1 dose) through Day 7. Participants will be treated with a single oral dose of 200 mg ETX0282 or placebo on the morning of Day 8. They will be confined to the Study Unit from Day -1 and discharged following collection of the 72-hour post Day 8 dose assessments (Day 11).
  Interventions: Drug: ETX0282; Drug: Placebo
- Part D: Cohort 12, ETX0282/Placebo plus Cefpodoxime Proxetil (Experimental): Part D of the study will explore the safety, tolerability, and PK of oral ETX0282 when administered as a single oral dose in combination with cefpodoxime proxetil tablets to healthy participants in a fed state. Participants will be treated with a single oral dose of 600 mg ETX0282 or placebo in a fed state on Day 1, with a single oral dose of 400 mg cefpodoxime proxetil in a fed state on Day 4, and with a single oral dose of 600 mg ETX0282 or placebo plus a single oral dose of 400 mg cefpodoxime proxetil dosed at the same time in a fed state on Day 7. They will be confined to the Study Unit from Day -1 and discharged following collection of the 72-hour post Day 7 dose assessments (Day 10).
  Interventions: Drug: ETX0282; Drug: Cefpodoxime proxetil; Drug: Placebo
- Part B (Food Effect): Cohort 14, 300 mg ETX0282/Placebo (Experimental): Part B of the study will explore the effect of food on oral ETX0282. Participants will be treated with a single oral dose of 300 mg ETX0282 or placebo (Day 1) while fasted and with a single oral dose of 300 mg ETX0282 or placebo (Day 4) with a high-fat meal. They will be confined to the Study Unit from Day -1 and discharged following collection of the 72-hour post fed state dose assessments (Day 7).
  Interventions: Drug: ETX0282; Drug: Placebo
- Part G: Cohort 17, 300 mg ETX0282/Placebo (Experimental): Part G of the study will explore the tolerability and PK profile of oral ETX0282 when administered either as a single dose (i.e., 300 mg as a single dose) or in 4 equal, divided doses over a 6 hour period (i.e., 75 mg every 2 hours for 4 doses [a 300 mg total dose]) when administered in a fasted state. Participants will receive the 2 treatments in a cross-over design according to one of 2 randomized sequences: AB or BA. Treatment A: 0 hours, 4 × 75 mg ETX0282/placebo; 2, 4, and 6 hours, 1 × 75 mg placebo. Treatment B: 0 hours, 1 × 75 mg ETX0282/placebo and 3 × 75 mg placebo; 2, 4, and 6 hours, 1 × 75 mg ETX0282/placebo. Participants will be confined to the Study Unit from Day -1 and discharged following collection of the 24 hours post Day 4 dose assessments (Day 5).
  Interventions: Drug: ETX0282; Drug: Placebo

INTERVENTIONS:
Drug: ETX0282 — Oral Gelatin capsules
Drug: Cefpodoxime proxetil — Oral tablets
  Arms: Part D: Cohort 12, ETX0282/Placebo plus Cefpodoxime Proxetil
Drug: Placebo — Oral Gelatin capsules

SUMMARY:
This research project is being conducted to investigate the safety, tolerability, and pharmacokinetics (PK) of a single ascending dose (SAD) and multiple ascending doses (MAD) of oral ETX0282 when administered alone and in combination with cefpodoxime proxetil in healthy adult participants.

DETAILED DESCRIPTION:
This Phase 1, single-center, double-blind, randomized, placebo-controlled study will be conducted to:

* Determine the safety and tolerability of oral ETX0282 when administered as a SAD and MAD to healthy participants;
* Determine the safety and tolerability of oral ETX0282 when administered as a single oral dose in combination with cefpodoxime proxetil to healthy participants;
* Characterize the PK in plasma and in urine of ETX0282 and ETX1317 following administration of single and multiple oral doses of ETX0282 in healthy participants; and
* Determine the PK profile in plasma and in urine of ETX0282 and ETX1317 and of cefpodoxime proxetil and cefpodoxime following administration of single oral doses of ETX0282 and cefpodoxime proxetil alone and when ETX0282 is co-administered with cefpodoxime proxetil at the same time as single oral doses in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 55 years (inclusive) for all participants except for those in Cohort 6 (in Part A); for Cohort 6, only participants aged ≥ 65 years will be enrolled.
* Be in general good health without clinically significant medical history
* Provide voluntary written informed consent prior to any study procedures and are willing and able to comply with the prescribed treatment protocol and evaluations
* Body mass index (BMI) ≥18.0 kilograms per meters squared (kg/m^2) and ≤32.0 kg/m^2
* Clinical laboratory values within the normal limits as defined by the clinical laboratory, unless the Principal Investigator decides that out-of-range values are not clinically significant
* Negative screen for drugs of abuse, alcohol, hepatitis B surface antigen, hepatitis C virus antibody, and human immunodeficiency virus at Screening; and drugs of abuse, alcohol predose on Day -1
* Female participants must be of non-childbearing potential (postmenopausal or with evidence of tubal ligation) or using a medically acceptable (highly effective method) contraceptive regimen and must have a negative pregnancy test at Screening (serum) and on Day -1 (urine) prior to study drug dosing. Male participants must be surgically sterile or using a medically acceptable contraceptive regimen. Men should not donate sperm during the study or for 90 days after the final dose of study medication.

Exclusion Criteria:

* History of any moderate or severe hypersensitivity or allergic reaction to any β-lactam antimicrobial (e.g., penicillin or cephalosporin)
* History of hypersensitivity or severe allergic reaction of any type to medications, bee stings, food, or environmental factors. A severe allergic reaction is defined as any of the following: anaphylaxis, urticaria, or angioedema.
* Use of prescription or over-the-counter medications within 7 days of investigational product administration, with the exception of contraceptive medications, paracetamol, oral non-steroidal anti-inflammatory agents, topical over-the-counter preparations, and routine vitamins (if they do not exceed an intake of 20 to 600 times the recommended daily dose), unless agreed as non-clinically relevant by the Principal Investigator and Sponsor
* Participation in an investigational drug or device study within 30 days before study drug dosing, i.e., there were at least 30 days between the last dose in a prior study and dose administration in this study
* Current smoker or difficulty abstaining from smoking for the duration of study confinement
* History of major organ dysfunction
* Infection or any serious underlying medical condition that would impair the participant from receiving study drug
* History of excessive alcohol intake (more than 4 standard drinks daily, on average) or use of recreational drugs within the last 3 months
* Standard donation of blood within 30 days of the study
* Concomitant disease or condition, including laboratory abnormality, which could interfere with the conduct of the study or which would, in the opinion of the Investigator, pose an unacceptable risk to the participant in this study
* Anticipated need for surgery or hospitalization during the study
* Surgery within 30 days before study enrolment
* Unwillingness or inability to comply with the study protocol for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with any non-serious adverse event | Up to 14 days after the last dose of study drug (Study Day [SD] 210)
Number of participants with any serious adverse event | Up to 14 days after the last dose of study drug (SD 210)
Number of participants with an adverse event of the indicated causality and severity | Up to 14 days after the last dose of study drug (SD 210)
Part A: Number of participants with abnormal, clinically significant hematology, clinical chemistry, and urinalysis laboratory values at the indicated time points | Screening (Day -1) up to Day 15±2 (Follow-up)
Part B: Number of participants with abnormal, clinically significant hematology, clinical chemistry, and urinalysis laboratory values at the indicated time points | Screening (Day -1; SD 44) up to Day 18±2 (SD 62±2; Follow-up)
Part C: Number of participants with abnormal, clinically significant hematology, clinical chemistry, and urinalysis laboratory values at the indicated time points | Screening (Day -1; SD 91) up to Day 22±2 (SD 113±2; Follow-up)
Part D: Number of participants with abnormal, clinically significant hematology, clinical chemistry, and urinalysis laboratory values at the indicated time points | Screening (Day -1; SD 142) up to Day 21±2 (SD 163±2; Follow-up)
Part G: Number of participants with abnormal, clinically significant hematology, clinical chemistry, and urinalysis laboratory values at the indicated time points | Screening (Day -1; SD 192) up to Day 18±2 (SD 210±2; Follow-up)
Part A: Number of participants with abnormal, clinically significant vital sign values at the indicated time points | Screening (Day -1) up to Day 15±2 (Follow-up)
Part B: Number of participants with abnormal, clinically significant vital sign values at the indicated time points | Screening (Day -1; SD 44) up to Day 18±2 (SD 62±2; Follow-up)
Part C: Number of participants with abnormal, clinically significant vital sign values at the indicated time points | Screening (Day -1; SD 91) up to Day 22±2 (SD 113±2; Follow-up)
Part D: Number of participants with abnormal, clinically significant vital sign values at the indicated time points | Screening (Day -1; SD 142) up to Day 21±2 (SD 163±2; Follow-up)
Part G: Number of participants with abnormal, clinically significant vital sign values at the indicated time points | Screening (Day -1; SD 192) up to Day 18±2 (SD 210±2; Follow-up)
Part A: Number of participants with abnormal, clinically significant electrocardiogram values at the indicated time points | Screening (Day -1) up to Day 15±2 (Follow-up)
Part B: Number of participants with abnormal, clinically significant electrocardiogram values at the indicated time points | Screening (Day -1; SD 44) up to Day 18±2 (SD 62±2; Follow-up)
Part C: Number of participants with abnormal, clinically significant electrocardiogram values at the indicated time points | Screening (Day -1; SD 91) up to Day 22±2 (SD 113±2; Follow-up)
Part D: Number of participants with abnormal, clinically significant electrocardiogram values at the indicated time points | Screening (Day -1; SD 142) up to Day 21±2 (SD 163±2; Follow-up)
Part G: Number of participants with abnormal, clinically significant electrocardiogram values at the indicated time points | Screening (Day -1; SD 192) up to Day 18±2 (SD 210±2; Follow-up)
Part A: Mean peak plasma concentration (Cmax) of ETX0282 and ETX1317 in blood in Cohorts 1 to 5 | Predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 (Day 1), 24 (Day 2), 48 (Day 3), and 72 (Day 4) hours postdose
Part A: Mean plasma concentration at time t (Ct) of ETX0282 and ETX1317 in blood in Cohorts 1 to 5 | Predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 (Day 1), 24 (Day 2), 48 (Day 3), and 72 (Day 4) hours postdose
Part A: Mean time to peak plasma concentration (Tmax) of ETX0282 and ETX1317 in blood in Cohorts 1 to 5 | Predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 (Day 1), 24 (Day 2), 48 (Day 3), and 72 (Day 4) hours postdose
Part A: Mean area under the concentration-time curve from time 0 to 24 hours (AUC0-24) of ETX0282 and ETX1317 in blood in Cohorts 1 to 5 | Predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 (Day 1), and 24 (Day 2) hours postdose
Part A: Mean area under the concentration-time curve from time 0 to the last time point evaluated (AUC0-t) of ETX0282 and ETX1317 in blood in Cohorts 1 to 5 | Predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 (Day 1), 24 (Day 2), 48 (Day 3), and 72 (Day 4) hours postdose
Part A: Mean area under the concentration-time curve from time 0 and extrapolated to infinity (AUC0-∞) of ETX0282 and ETX1317 in blood in Cohorts 1 to 5 | Predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 (Day 1), 24 (Day 2), 48 (Day 3), and 72 (Day 4) hours postdose
Part A: Mean elimination rate constant (Kel) of ETX0282 and ETX1317 in blood in Cohorts 1 to 5 | Predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 (Day 1), 24 (Day 2), 48 (Day 3), and 72 (Day 4) hours postdose
Part A: Mean elimination half-life (t½) of ETX0282 and ETX1317 in blood in Cohorts 1 to 5 | Predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 (Day 1), 24 (Day 2), 48 (Day 3), and 72 (Day 4) hours postdose
Part A: Mean clearance (CL) of ETX0282 and ETX1317 in blood in Cohorts 1 to 5 | Predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 (Day 1), 24 (Day 2), 48 (Day 3), and 72 (Day 4) hours postdose
Part A: Mean volume of distribution (Vdss) of ETX0282 and ETX1317 in blood in Cohorts 1 to 5 | Predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 (Day 1), 24 (Day 2), 48 (Day 3), and 72 (Day 4) hours postdose
Part A: Mean cumulative excretion of unchanged ETX0282 and ETX1317 in urine (Ae) in Cohorts 1 to 5 | Prior to dosing (-6 to 0 hours; Day 1); 0 to 8 (Day 1), 8 to 24 (Day 2), 24 to 48 (Day 3), and 48 to 72 (Day 4) hours postdose
Part A: Mean urinary clearance (CLR) of ETX0282 and ETX1317 in Cohorts 1 to 5 | Prior to dosing (-6 to 0 hours; Day 1); 0 to 8 (Day 1), 8 to 24 (Day 2), 24 to 48 (Day 3), and 48 to 72 (Day 4) hours postdose
Part A: Mean fraction of the administered dose of ETX0282 and ETX1317 that is excreted unchanged in the urine (fe) in Cohorts 1 to 5 | Prior to dosing (-6 to 0 hours; Day 1); 0 to 8 (Day 1), 8 to 24 (Day 2), 24 to 48 (Day 3), and 48 to 72 (Day 4) hours postdose
Part A: Mean dose proportionality of ETX0282 and ETX1317 in Cohorts 1 to 5 | Predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 (Day 1), 24 (Day 2), 48 (Day 3), and 72 (Day 4) hours postdose
Part C: Mean Cmax of ETX0282 and ETX1317 in blood | Days 1-3, 5, and 8 (SDs 92-94, 96, and 99): predose (30 min); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours post first dose; at troughs of Days 3, 5, and 8 (SDs 94, 96, and 99); at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post last dose
  min, minutes
Part C: Mean Ct of ETX0282 and ETX1317 in blood | Days 1-3, 5, and 8 (SDs 92-94, 96, and 99): predose (30 min); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours post first dose; at troughs of Days 3, 5, and 8 (SDs 94, 96, and 99); at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post last dose
Part C: Mean Tmax of ETX0282 and ETX1317 in blood | Days 1-3, 5, and 8 (SDs 92-94, 96, and 99): predose (30 min); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours post first dose; at troughs of Days 3, 5, and 8 (SDs 94, 96, and 99); at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post last dose
Part C: Mean AUC0-24 of ETX0282 and ETX1317 in blood | Days 1-3, 5, and 8 (SDs 92-94, 96, and 99): predose (30 min); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours post first dose; at troughs of Days 3, 5, and 8 (SDs 94, 96, and 99); at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post last dose
Part C: Mean AUC0-t of ETX0282 and ETX1317 in blood | Days 1-3, 5, and 8 (SDs 92-94, 96, and 99): predose (30 min); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours post first dose; at troughs of Days 3, 5, and 8 (SDs 94, 96, and 99); at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post last dose
Part C: Mean AUC0-∞ of ETX0282 and ETX1317 in blood | Days 1-3, 5, and 8 (SDs 92-94, 96, and 99): predose (30 min); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours post first dose; at troughs of Days 3, 5, and 8 (SDs 94, 96, and 99); at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post last dose
Part C: Mean AUC from time 0 to the end of the dosing period (AUC0-tau) of ETX0282 and ETX1317 in blood | Days 1-3, 5, and 8 (SDs 92-94, 96, and 99): predose (30 min); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours post first dose; at troughs of Days 3, 5, and 8 (SDs 94, 96, and 99); at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post last dose
Part C: Mean accumulation ratio (R0) of ETX0282 and ETX1317 in blood | Days 1-3, 5, and 8 (SDs 92-94, 96, and 99): predose (30 min); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours post first dose; at troughs of Days 3, 5, and 8 (SDs 94, 96, and 99); at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post last dose
Part C: Mean Kel of ETX0282 and ETX1317 in blood | Days 1-3, 5, and 8 (SDs 92-94, 96, and 99): predose (30 min); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours post first dose; at troughs of Days 3, 5, and 8 (SDs 94, 96, and 99); at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post last dose
Part C: Mean t½ of ETX0282 and ETX1317 in blood | Days 1-3, 5, and 8 (SDs 92-94, 96, and 99): predose (30 min); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours post first dose; at troughs of Days 3, 5, and 8 (SDs 94, 96, and 99); at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post last dose
Part C: Mean CL of ETX0282 and ETX1317 in blood | Days 1-3, 5, and 8 (SDs 92-94, 96, and 99): predose (30 min); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours post first dose; at troughs of Days 3, 5, and 8 (SDs 94, 96, and 99); at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post last dose
Part C: Mean Vdss of ETX0282 and ETX1317 in blood | Days 1-3, 5, and 8 (SDs 92-94, 96, and 99): predose (30 min); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours post first dose; at troughs of Days 3, 5, and 8 (SDs 94, 96, and 99); at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post last dose
Part C: Mean Ae of ETX0282 and ETX1317 | Days 1-4 and 8-11 (SDs 92-95 and 99-102): prior to dosing (-6 to 0 hours; first and last doses) and at 0-8, 8-24, 24-48, and 48-72 hours post first and last dose
Part C: Mean CLR of ETX0282 and ETX1317 | Days 1-4 and 8-11 (SDs 92-95 and 99-102): prior to dosing (-6 to 0 hours; first and last doses) and at 0-8, 8-24, 24-48, and 48-72 hours post first and last dose
Part C: Mean fe of ETX0282 and ETX1317 | Days 1-4 and 8-11 (SDs 92-95 and 99-102): prior to dosing (-6 to 0 hours; first and last doses) and at 0-8, 8-24, 24-48, and 48-72 hours post first and last dose
Part C: Mean dose proportionality of ETX0282 and ETX1317 | Days 1-3, 5, and 8 (SDs 92-94, 96, and 99): predose (30 min); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours post first dose; at troughs of Days 3, 5, and 8 (SDs 94, 96, and 99); at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, and 12 hours post last dose
Part D: Mean Cmax of ETX0282 and ETX1317 in blood | Days 1-10 (SDs 143-152): predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours postdose
Part D: Mean Ct of ETX0282 and ETX1317 in blood | Days 1-10 (SDs 143-152): predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours postdose
Part D: Mean Tmax of ETX0282 and ETX1317 in blood | Days 1-10 (SDs 143-152): predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours postdose
Part D: Mean AUC0-24 of ETX0282 and ETX1317 in blood | Days 1-10 (SDs 143-152): predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours postdose
Part D: Mean AUC0-t of ETX0282 and ETX1317 in blood | Days 1-10 (SDs 143-152): predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours postdose
Part D: Mean AUC0-∞ of ETX0282 and ETX1317 in blood | Days 1-10 (SDs 143-152): predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours postdose
Part D: Mean Kel of ETX0282 and ETX1317 in blood | Days 1-10 (SDs 143-152): predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours postdose
Part D: Mean t½ of ETX0282 and ETX1317 in blood | Days 1-10 (SDs 143-152): predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours postdose
Part D: Mean CL of ETX0282 and ETX1317 in blood | Days 1-10 (SDs 143-152): predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours postdose
Part D: Mean Vdss of ETX0282 and ETX1317 in blood | Days 1-10 (SDs 143-152): predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours postdose
Part D: Mean Ae of ETX0282 and ETX1317 | Days 1-10 (SDs 143-152): prior to dosing (-6 to 0 hours) and at 0-8, 8-24, 24-48, and 48-72 hours postdose
Part D: Mean CLR of ETX0282 and ETX1317 | Days 1-10 (SDs 143-152): prior to dosing (-6 to 0 hours) and at 0-8, 8-24, 24-48, and 48-72 hours postdose
Part D: Mean fe of ETX0282 and ETX1317 | Days 1-10 (SDs 143-152): prior to dosing (-6 to 0 hours) and at 0-8, 8-24, 24-48, and 48-72 hours postdose
Part D: Mean dose proportionality of ETX0282 and ETX1317 | Days 1-10 (SDs 143-152): predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours postdose
Part D: Mean Cmax of cefpodoxime proxetil and cefpodoxime following administration of cefpodoxime proxetil as a single oral dose either alone or in combination with ETX0282 | Days 1-10 (SDs 143-152): predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours postdose
Part D: Mean Ct of cefpodoxime proxetil and cefpodoxime following administration of cefpodoxime proxetil as a single oral dose either alone or in combination with ETX0282 | Days 1-10 (SDs 143-152): predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours postdose
Part D: Mean Tmax of cefpodoxime proxetil and cefpodoxime following administration of cefpodoxime proxetil as a single oral dose either alone or in combination with ETX0282 | Days 1-10 (SDs 143-152): predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours postdose
Part D: Mean AUC0-24 of cefpodoxime proxetil and cefpodoxime following administration of cefpodoxime proxetil as a single oral dose either alone or in combination with ETX0282 | Days 1-10 (SDs 143-152): predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, and 24 hours postdose
Part D: Mean AUC0-t of cefpodoxime proxetil and cefpodoxime following administration of cefpodoxime proxetil as a single oral dose either alone or in combination with ETX0282 | Days 1-10 (SDs 143-152): predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours postdose
Part D: Mean AUC0-∞ of cefpodoxime proxetil and cefpodoxime following administration of cefpodoxime proxetil as a single oral dose either alone or in combination with ETX0282 | Days 1-10 (SDs 143-152): predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours postdose
Part D: Mean Kel of cefpodoxime proxetil and cefpodoxime following administration of cefpodoxime proxetil as a single oral dose either alone or in combination with ETX0282 | Days 1-10 (SDs 143-152): predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours postdose
Part D: Mean t½ of cefpodoxime proxetil and cefpodoxime following administration of cefpodoxime proxetil as a single oral dose either alone or in combination with ETX0282 | Days 1-10 (SDs 143-152): predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours postdose
Part D: Mean CL of cefpodoxime proxetil and cefpodoxime following administration of cefpodoxime proxetil as a single oral dose either alone or in combination with ETX0282 | Days 1-10 (SDs 143-152): predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours postdose
Part D: Mean Vdss of cefpodoxime proxetil and cefpodoxime following administration of cefpodoxime proxetil as a single oral dose either alone or in combination with ETX0282 | Days 1-10 (SDs 143-152): predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours postdose
Part D: Mean Ae of cefpodoxime proxetil and cefpodoxime following administration of cefpodoxime proxetil as a single oral dose either alone or in combination with ETX0282 | Days 1-10 (SDs 143-152): prior to dosing (-6 to 0 hours) and at 0-8, 8-24, 24-48, and 48-72 hours postdose
Part D: Mean CLR of cefpodoxime proxetil and cefpodoxime following administration of cefpodoxime proxetil as a single oral dose either alone or in combination with ETX0282 | Days 1-10 (SDs 143-152): prior to dosing (-6 to 0 hours) and at 0-8, 8-24, 24-48, and 48-72 hours postdose
Part D: Mean fe of cefpodoxime proxetil and cefpodoxime following administration of cefpodoxime proxetil as a single oral dose either alone or in combination with ETX0282 | Days 1-10 (SDs 143-152): prior to dosing (-6 to 0 hours) and at 0-8, 8-24, 24-48, and 48-72 hours postdose
Part D: Mean dose proportionality of cefpodoxime proxetil and cefpodoxime following administration of cefpodoxime proxetil as a single oral dose either alone or in combination with ETX0282 | Days 1-10 (SDs 143-152): predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 48, and 72 hours postdose
Part G: Mean Cmax of ETX0282 and ETX1317 in blood | Days 1 and 4 (SDs 193 and 196): 30 minutes predose; 0.25, 0.5, 0.75, 1, 1.5, 2 (predose prior to subsequent dose), 2.5, 3, 4 (predose prior to subsequent dose), 7, 8, 12, and 16 hours postdose. Days 2 and 5 (SDs 194 and 197): 24 hours postdose
Part G: Mean Ct of ETX0282 and ETX1317 in blood | Days 1 and 4 (SDs 193 and 196): 30 minutes predose; 0.25, 0.5, 0.75, 1, 1.5, 2 (predose prior to subsequent dose), 2.5, 3, 4 (predose prior to subsequent dose), 7, 8, 12, and 16 hours postdose. Days 2 and 5 (SDs 194 and 197): 24 hours postdose
Part G: Mean Tmax of ETX0282 and ETX1317 in blood | Days 1 and 4 (SDs 193 and 196): 30 minutes predose; 0.25, 0.5, 0.75, 1, 1.5, 2 (predose prior to subsequent dose), 2.5, 3, 4 (predose prior to subsequent dose), 7, 8, 12, and 16 hours postdose. Days 2 and 5 (SDs 194 and 197): 24 hours postdose
Part G: Mean AUC0-24 of ETX0282 and ETX1317 in blood | Days 1 and 4 (SDs 193 and 196): 30 minutes predose; 0.25, 0.5, 0.75, 1, 1.5, 2 (predose prior to subsequent dose), 2.5, 3, 4 (predose prior to subsequent dose), 7, 8, 12, and 16 hours postdose. Days 2 and 5 (SDs 194 and 197): 24 hours postdose
Part G: Mean AUC0-t of ETX0282 and ETX1317 in blood | Days 1 and 4 (SDs 193 and 196): 30 minutes predose; 0.25, 0.5, 0.75, 1, 1.5, 2 (predose prior to subsequent dose), 2.5, 3, 4 (predose prior to subsequent dose), 7, 8, 12, and 16 hours postdose. Days 2 and 5 (SDs 194 and 197): 24 hours postdose
Part G: Mean AUC0-∞ of ETX0282 and ETX1317 in blood | Days 1 and 4 (SDs 193 and 196): 30 minutes predose; 0.25, 0.5, 0.75, 1, 1.5, 2 (predose prior to subsequent dose), 2.5, 3, 4 (predose prior to subsequent dose), 7, 8, 12, and 16 hours postdose. Days 2 and 5 (SDs 194 and 197): 24 hours postdose
Part G: Mean AUC0-tau of ETX0282 and ETX1317 in blood | Days 1 and 4 (SDs 193 and 196): 30 minutes predose; 0.25, 0.5, 0.75, 1, 1.5, 2 (predose prior to subsequent dose), 2.5, 3, 4 (predose prior to subsequent dose), 7, 8, 12, and 16 hours postdose. Days 2 and 5 (SDs 194 and 197): 24 hours postdose
Part G: Mean R0 of ETX0282 and ETX1317 in blood | Days 1 and 4 (SDs 193 and 196): 30 minutes predose; 0.25, 0.5, 0.75, 1, 1.5, 2 (predose prior to subsequent dose), 2.5, 3, 4 (predose prior to subsequent dose), 7, 8, 12, and 16 hours postdose. Days 2 and 5 (SDs 194 and 197): 24 hours postdose
Part G: Mean Kel of ETX0282 and ETX1317 in blood | Days 1 and 4 (SDs 193 and 196): 30 minutes predose; 0.25, 0.5, 0.75, 1, 1.5, 2 (predose prior to subsequent dose), 2.5, 3, 4 (predose prior to subsequent dose), 7, 8, 12, and 16 hours postdose. Days 2 and 5 (SDs 194 and 197): 24 hours postdose
Part G: Mean t½ of ETX0282 and ETX1317 in blood | Days 1 and 4 (SDs 193 and 196): 30 minutes predose; 0.25, 0.5, 0.75, 1, 1.5, 2 (predose prior to subsequent dose), 2.5, 3, 4 (predose prior to subsequent dose), 7, 8, 12, and 16 hours postdose. Days 2 and 5 (SDs 194 and 197): 24 hours postdose
Part G: Mean CL of ETX0282 and ETX1317 in blood | Days 1 and 4 (SDs 193 and 196): 30 minutes predose; 0.25, 0.5, 0.75, 1, 1.5, 2 (predose prior to subsequent dose), 2.5, 3, 4 (predose prior to subsequent dose), 7, 8, 12, and 16 hours postdose. Days 2 and 5 (SDs 194 and 197): 24 hours postdose
Part G: Mean Vdss of ETX0282 and ETX1317 in blood | Days 1 and 4 (SDs 193 and 196): 30 minutes predose; 0.25, 0.5, 0.75, 1, 1.5, 2 (predose prior to subsequent dose), 2.5, 3, 4 (predose prior to subsequent dose), 7, 8, 12, and 16 hours postdose. Days 2 and 5 (SDs 194 and 197): 24 hours postdose
Part G: Mean Ae of ETX0282 and ETX1317 | Days 1 and 4 (SDs 193 and 196): 30 minutes predose; 0.25, 0.5, 0.75, 1, 1.5, 2 (predose prior to subsequent dose), 2.5, 3, 4 (predose prior to subsequent dose), 7, 8, 12, and 16 hours postdose. Days 2 and 5 (SDs 194 and 197): 24 hours postdose
Part G: Mean CLR of ETX0282 and ETX1317 | Days 1 and 4 (SDs 193 and 196): 30 minutes predose; 0.25, 0.5, 0.75, 1, 1.5, 2 (predose prior to subsequent dose), 2.5, 3, 4 (predose prior to subsequent dose), 7, 8, 12, and 16 hours postdose. Days 2 and 5 (SDs 194 and 197): 24 hours postdose
Part G: Mean fe of ETX0282 and ETX1317 | Days 1 and 4 (SDs 193 and 196): 30 minutes predose; 0.25, 0.5, 0.75, 1, 1.5, 2 (predose prior to subsequent dose), 2.5, 3, 4 (predose prior to subsequent dose), 7, 8, 12, and 16 hours postdose. Days 2 and 5 (SDs 194 and 197): 24 hours postdose
Part G: Mean dose proportionality of ETX0282 and ETX1317 | Days 1 and 4 (SDs 193 and 196): 30 minutes predose; 0.25, 0.5, 0.75, 1, 1.5, 2 (predose prior to subsequent dose), 2.5, 3, 4 (predose prior to subsequent dose), 7, 8, 12, and 16 hours postdose. Days 2 and 5 (SDs 194 and 197): 24 hours postdose

SECONDARY OUTCOMES:
Number of elderly participants with any non-serious adverse event | Up to 14 days after the last dose of study drug (SD 210)
Number of elderly participants with any serious adverse event | Up to 14 days after the last dose of study drug (SD 210)
Number of elderly participants with an adverse event of the indicated causality and severity | Up to 14 days after the last dose of study drug (SD 210)
Part A: Number of elderly participants with abnormal, clinically significant hematology, clinical chemistry, and urinalysis laboratory values at the indicated time points | Screening (Day -1); Days 2, 3, 4, 7, and 15±2 (Follow-up)
Part A: Number of elderly participants with abnormal, clinically significant vital sign values at the indicated time points | Screening (Day -1); Days 2, 3, 4, 7, and 15±2 (Follow-up)
Part A: Number of elderly participants with abnormal, clinically significant electrocardiogram values at the indicated time points | Screening (Day -1); Days 1-7; Day 15±2 (Follow-up)
Number of participants who received concomitant medications | Up to 14 days after the last dose of study drug (SD 210)
  Concomitant medications will be coded using the World Health Organization Drug Dictionary. The incidence of participants taking each medication by Anatomical Therapeutic Chemical second and fourth level categories (pharmacological or therapeutic group) will be presented.
Part A: Mean Cmax of ETX0282 and ETX1317 in blood of elderly participants (Cohort 6) | Predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 (Day 1), 24 (Day 2), 48 (Day 3), and 72 (Day 4) hours postdose
Part A: Mean Ct of ETX0282 and ETX1317 in blood of elderly participants (Cohort 6) | Predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 (Day 1), 24 (Day 2), 48 (Day 3), and 72 (Day 4) hours postdose
Part A: Mean Tmax of ETX0282 and ETX1317 in blood of elderly participants (Cohort 6) | Predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 (Day 1), 24 (Day 2), 48 (Day 3), and 72 (Day 4) hours postdose
Part A: Mean AUC0-24 of ETX0282 and ETX1317 in blood of elderly participants (Cohort 6) | Predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 (Day 1), and 24 (Day 2) hours postdose
Part A: Mean AUC0-t of ETX0282 and ETX1317 in blood of elderly participants (Cohort 6) | Predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 (Day 1), 24 (Day 2), 48 (Day 3), and 72 (Day 4) hours postdose
Part A: Mean AUC0-∞ of ETX0282 and ETX1317 in blood of elderly participants (Cohort 6) | Predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 (Day 1), 24 (Day 2), 48 (Day 3), and 72 (Day 4) hours postdose
Part A: Mean Kel of ETX0282 and ETX1317 in blood of elderly participants (Cohort 6) | Predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 (Day 1), 24 (Day 2), 48 (Day 3), and 72 (Day 4) hours postdose
Part A: Mean t½ of ETX0282 and ETX1317 in blood of elderly participants (Cohort 6) | Predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 (Day 1), 24 (Day 2), 48 (Day 3), and 72 (Day 4) hours postdose
Part A: Mean CL of ETX0282 and ETX1317 in blood of elderly participants (Cohort 6) | Predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 (Day 1), 24 (Day 2), 48 (Day 3), and 72 (Day 4) hours postdose
Part A: Mean Vdss of ETX0282 and ETX1317 in blood of elderly participants (Cohort 6) | Predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 (Day 1), 24 (Day 2), 48 (Day 3), and 72 (Day 4) hours postdose
Part A: Mean Ae of ETX0282 and ETX1317 for elderly participants (Cohort 6) | Prior to dosing (-6 to 0 hours; Day 1); 0 to 8 (Day 1), 8 to 24 (Day 2), 24 to 48 (Day 3), and 48 to 72 (Day 4) hours postdose
Part A: Mean CLR of ETX0282 and ETX1317 in urine for elderly participants (Cohort 6) | Prior to dosing (-6 to 0 hours; Day 1); 0 to 8 (Day 1), 8 to 24 (Day 2), 24 to 48 (Day 3), and 48 to 72 (Day 4) hours postdose
Part A: Mean fe of ETX0282 and ETX1317 for elderly participants (Cohort 6) | Prior to dosing (-6 to 0 hours; Day 1); 0 to 8 (Day 1), 8 to 24 (Day 2), 24 to 48 (Day 3), and 48 to 72 (Day 4) hours postdose
Part A: Mean dose proportionality of ETX0282 and ETX1317 for elderly participants (Cohort 6) | Predose (0); 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 (Day 1), 24 (Day 2), 48 (Day 3), and 72 (Day 4) hours postdose
Part B: Mean Cmax of ETX0282 and ETX1317 in blood | Days 1-7 (SDs 45-51): predose (0), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 16, 24, 48, and 72 hours postdose
Part B: Mean Ct of ETX0282 and ETX1317 in blood | Days 1-7 (SDs 45-51): predose (0), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 16, 24, 48, and 72 hours postdose
Part B: Mean Tmax of ETX0282 and ETX1317 in blood | Days 1-7 (SDs 45-51): predose (0), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 16, 24, 48, and 72 hours postdose
Part B: Mean AUC0-24 of ETX0282 and ETX1317 in blood | Days 1-7 (SDs 45-51): predose (0), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 16, and 24 hours postdose
Part B: Mean AUC0-t of ETX0282 and ETX1317 in blood | Days 1-7 (SDs 45-51): predose (0), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 16, 24, 48, and 72 hours postdose
Part B: Mean AUC0-∞ of ETX0282 and ETX1317 in blood | Days 1-7 (SDs 45-51): predose (0), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 16, 24, 48, and 72 hours postdose
Part B: Mean Kel of ETX0282 and ETX1317 in blood | Days 1-7 (SDs 45-51): predose (0), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 16, 24, 48, and 72 hours postdose
Part B: Mean t½ of ETX0282 and ETX1317 in blood | Days 1-7 (SDs 45-51): predose (0), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 16, 24, 48, and 72 hours postdose
Part B: Mean CL of ETX0282 and ETX1317 in blood | Days 1-7 (SDs 45-51): predose (0), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 16, 24, 48, and 72 hours postdose
Part B: Mean Vdss of ETX0282 and ETX1317 in blood | Days 1-7 (SDs 45-51): predose (0), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 16, 24, 48, and 72 hours postdose
Part B: Mean Ae of ETX0282 and ETX1317 | Days 1-7 (SDs 45-51): prior to dosing (-6 to 0 hours) and at 0-8, 8-24, 24-48, and 48-72 hours postdose
Part B: Mean CLR of ETX0282 and ETX1317 | Days 1-7 (SDs 45-51): prior to dosing (-6 to 0 hours) and at 0-8, 8-24, 24-48, and 48-72 hours postdose
Part B: Mean fe of ETX0282 and ETX1317 | Days 1-7 (SDs 45-51): prior to dosing (-6 to 0 hours) and at 0-8, 8-24, 24-48, and 48-72 hours postdose
Part B: Mean dose proportionality of ETX0282 and ETX1317 | Days 1-7 (SDs 45-51): predose (0), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 8, 12, 16, 24, 48, and 72 hours postdose

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia